CLINICAL TRIAL: NCT00839475
Title: Investigational Study: Imaging the Uterine Cervix Using C30 Investigational Device
Brief Title: Investigation of the Uterine Cervix Using CervicalMD
Status: Completed | Type: Observational
Sponsor: STI-Medical Systems (Industry)
Responsible Party: Jody Oyama, Clinical Director, STI-Medical Systems,
Other Study IDs: 2008-1
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Colposcopy
Keywords: colposcopy; Cervical intraepithelial neoplasia; cervical cancer; cervical precancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — LEEP specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate the CervicalMD device's ability to collect digital imagery suitable for a colposcopy examination.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Negative Pregnancy test
* Abnormal Pap smear
* 18 years and older
* Presence of a cervix

Exclusion Criteria:

* Pregnant
* Absence of a cervix
* Less than 18 years old
* Male

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women identified with an abnormal Pap smear
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daron G Ferris, MD, Principal Investigator — Augusta University